CLINICAL TRIAL: NCT03727789
Title: A Single-Center Phase I Dose Escalation/Response Trial to Evaluate Safety, Tolerability, and Anti-Tumor Efficacy of Intra-Arterial CBL0137 for Patients With Advanced Extremity Melanoma or Sarcoma
Brief Title: CBL0137 in Treating Patients With Advanced Extremity Melanoma or Sarcoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Incuron (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 60017; NCI-2018-01928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 60017 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-10-12; First posted 2018-11-01 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Advanced Cutaneous Melanoma of the Extremity; Advanced Sarcoma of the Extremity; Clinical Stage III Cutaneous Melanoma AJCC v8; Clinical Stage IV Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IV Cutaneous Melanoma AJCC v8; Recurrent Cutaneous Melanoma of the Extremity; Recurrent Sarcoma of the Extremity; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IV Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8
MeSH Terms: interventions — CBLC137

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CBL0137) (Experimental): Patients receive FACT complex-targeting curaxin CBL0137 IA over 15 minutes.
  Interventions: Drug: FACT Complex-targeting Curaxin CBL0137

INTERVENTIONS:
Drug: FACT Complex-targeting Curaxin CBL0137 — Given IA
  Other Names: CBL0137

SUMMARY:
This phase I trial studies best dose and side effects of CBL0137 in treating patients with extremity melanoma or sarcoma that has spread to other places in the body. Drugs, such as CBL0137, may work by binding to tumor cell deoxyribonucleic acid (DNA) to stop the cell from growing further.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and examine the dose-limiting toxicities of intra-arterial facilitates chromatin transcription (FACT) complex-targeting curaxin CBL0137 (CBL0137) in patients with advanced extremity melanoma or sarcoma.

SECONDARY OBJECTIVES:

I. To assess the tumor response in advanced melanoma and sarcoma patients treated with intra-arterial administration of CBL0137.

II. To define both response in-field (area of the limb distal to the infusion point) and out-of-field (any area proximal to the infusion point) in patients treated with CBL0137 based intra-arterial infusion.

III. Assess the pharmacokinetics of CBL0137 in the study population pre-and post CBL0137 intraarterial infusion.

IV. Assess tumor protein expression profiles before and after treatment with CBL0137.

TERTIARY OBJECTIVES:

I. To assess if the proposed treatment has any effect on quality of life as measured by the Functional Assessment of Cancer Therapy ? Melanoma (assessment tool also applicable to sarcoma).

OUTLINE: This is a dose-escalation study of FACT complex-targeting curaxin CBL0137.

Patients receive FACT complex-targeting curaxin CBL0137 intra-arterially (IA) over 15 minutes.

After completion of study treatment, patients are followed up at 2, 6 and 12 weeks, every 3 months for 12 months, then at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a life expectancy of > 6 months.
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
* Patients either:

  * Must not have undergone any limb-directed treatment OR
  * Have undergone a previous Melphalan based regional therapy for which they did not have a complete response and, present with persistent, progressive, or recurrent disease.
* * NOTE: Patients with indeterminate staging must be reviewed by the Principal Investigator prior to registration.
* Patient must have had a washout period for at least 30 days or 5 half-lives from any prior chemotherapy, radioactive, or hormonal cancer therapy, or 4 weeks from any checkpoint inhibitors or other biologic (including TVEC), whichever is longer
* Patient must have histologically proven primary or recurrent extremity melanoma (stage IIIB, IIIC, or IV), or advanced extremity sarcoma not amenable to surgical resection

  * (American Joint Committee on Cancer [AJCC] melanoma staging must be documented in patient's medical record, as determined by computed tomography [CT] of the chest, abdomen and pelvis, within six weeks prior to administration of study drug;
  * Due to the heterogeneous nature of sarcoma, AJCC sarcoma staging is NOT required
* Patients with Stage IIIC disease must either have had regional lymph nodes previously removed or have stable or regressed disease on imaging from prior systemic therapy (defined as modified RECIST 1.1 SD, CR, or PR).

  * Stable or regressed disease must be present for at least the 2 months prior to IA CBL0137 and patient is no longer receiving systemic therapy (with the exception of immunotherapy) during this time period for melanoma.
  * Stable or regressed disease must be present for at least the 2 months prior to IA CBL0137 and patient is no longer receiving systemic therapy during this time period for sarcoma
* Patients with Stage IV disease must have had all distant disease resected at least 30 days prior to regional treatment, or exhibit stable or regressed disease .on imaging from prior systemic therapy (defined as modified RECIST 1.1 SD, CR, or PR).

  * Stable or regressed disease must be present for at least the 2 months prior to IA CBL0137 and patient is not receiving systemic therapy (with the exception of immunotherapy) during this time period for melanoma
  * Stable or regressed disease must be present for at least the 2 months prior to IA CBL0137 and patient is no longer receiving systemic therapy during this time period for sarcoma
* Melanoma or sarcoma patients who have stable or completely responded brain metastases from previous gamma knife surgery and/or systemic therapies are eligible.
* Patient's disease must be measurable by caliper or radiological method as defined in the modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
* Patient must have adequate bone marrow, liver and renal function as assessed by the following:
* Hemoglobin >= 9 g/dL.
* White blood count (WBC) of >= 3000 m^3.
* Absolute neutrophil count (ANC) >= 1,500/mm^3.
* Platelet count >= 100,000/mm^3.
* Total bilirubin =< 1.5 x upper limit of normal (ULN).
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x the ULN.
* Creatinine clearance (CrCl) > 45 mL/minute.
* Patient must have a palpable femoral/radial pulse in the affected extremity.
* Patients must have recovered from adverse events from previously administered agents (<=grade 2) prior to first study drug administration
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to read and understand English and the ability to complete paper and/or electronic survey assessments.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Cardiac disease: Congestive heart failure > Class II New York Heart Association (NYHA). Patients must not have unstable angina (angina symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months
* Males with mean QTcF values of >450 msec and females with QTcF values of >470 msec, patients who are known to have congenital prolonged QT syndromes, or patients who are on medications known to cause prolonged QT intervals on ECG.
* Use of drugs known to prolong QT.
* Patients with known hypersensitivity to any of the components of CBL0137.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Thrombotic ((excluding prior catheter-related thrombus that has been adequately treated) or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Patients with symptoms or signs of vascular insufficiency. Specifically, patients with any history of blood clots (excluding prior catheter-related thrombus that has been adequately treated) or lifestyle altering ischemic peripheral vascular disease will be excluded.
* Evidence or history of bleeding diathesis or coagulopathy.
* Patients with known heparin induced thrombocytopenia.
* Untreated or growing brain metastasis: Patients with neurological symptoms must undergo a CT scan/magnetic resonance imaging (MRI) of the brain to exclude untreated or growing brain metastasis.
* Known human immunodeficiency virus (HIV) infection or active hepatitis B or C.
* Active clinically serious infection > Common Terminology Criteria for Adverse Events (CTCAE) Grade 2.
* Serious non-healing wound, ulcer, or bone fracture.
* Major surgery or significant traumatic injury within 30 days of planned intra-arterial infusion.
* Current treatment or, treatment within the previous 24 months, for another non-melanoma or sarcoma malignancy.
* Patients who have already received 2 prior infusions of CBL0137.
* Pregnant or nursing female participants.
* Psychiatric conditions or diminished capacity that could compromise the giving of informed consent, or interfere with study compliance.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the Investigator?s opinion deems the participant an unsuitable candidate to receive study drug.
* Received an investigational agent within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) defined based on the rate of drug-related grade 3-5 adverse events assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events version (CTCAE) (v.) 5. | Up to 24 months
  The frequency of toxicities will be tabulated by grade across all dose levels. The frequency of toxicities will also be tabulated for the dose estimated to be the maximum tolerated dose.

SECONDARY OUTCOMES:
Tumor response as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 modified for cutaneous, out-of-field, and deeper lesions | Up to 24 months
  Responses will be tabulated, and complete response rate will be estimated with its exact 80% confidence interval.
Duration of tumor response (both in the field of infusion therapy and out-of-field) assessed by RECIST 1.1 | Up to 24 months
Duration of regional progression free survival (PFS) assessed by RECIST 1.1 | Up to 24 months
Overall PFS assessed by RECIST 1.1 | Up to 24 months
Incidence and type of adverse events assessed using NCI CTCAE v.5 | Up to 24 months
Incidence of Adverse Events | Baseline up to 24 months
  Changes in clinical laboratory values while receiving CBL0137
Incidence of Adverse events | At pre- and post-intraarterial infusion assessed up to 24 months
  Drug safety
Tumor levels of p53^Ser392 and HSP70 assessed by enzyme-linked immunosorbent assay (ELISA) | Up to 24 months

OTHER OUTCOMES:
Quality of life (QOL) measured using the Functional Assessment of Cancer Therapy - Melanoma (FACT-M v.4) and the associated Melanoma Cancer subscale (MCS) | Up to 24 months
  Median and range baseline subscale and total QOL scores, as well as single item scores, will be presented, followed by mean change scores for subscales, the total scale and single items, compared between different study intervention groups.
Quality of life (QOL) measured using the associated Melanoma Cancer subscale (MCS) | Up to 24 months
  Median and range baseline subscale and total QOL scores, as well as single item scores, will be presented, followed by mean change scores for subscales, the total scale and single items, compared between different study intervention groups.
Melanoma-related symptoms measured using the FACT-M v.4 | Up to 24 months
Melanoma-related symptoms measured using the associated Melanoma Cancer Subscale | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Skitzki, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States